CLINICAL TRIAL: NCT07183267
Title: Reducing rAdiation aDverse Effects of dermatitIs and mucosAl inflammatioN Using Red Light Therapy
Brief Title: Using Red Light Therapy to Ease Skin Side Effects and Mouth Side Effects, in Children and Young People Aged 0 to 16 Years Old, Receiving Radiotherapy
Acronym: RADIANT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CFTSp248
Record Dates: First submitted 2025-08-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Radio Dermatitis; Mucositis Oral; Oesophagitis
Keywords: Paediatric skin toxicity; paediatric oral mucositis; paediatric proton therapy; paediatric radiotherapy; paediatric photon therapy
MeSH Terms: conditions — Stomatitis; Esophagitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photobiomodulation (Experimental): Participants will received a daily treatment of photobiomodulation via a LED photobiomodulation device alongside their proton or photon treatment fraction. The photobiomodulation will be administered to the skin in the site of the patients proton or photon therapy treatment area.
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Participants will received a daily treatment of photobiomodulation via a LED photobiomodulation device alongside their proton or photon treatment fraction. The photobiomodulation will be administered to the skin in the site of the patients proton or photon therapy treatment area.
  Other Names: Red light therapy; LED light therapy

SUMMARY:
The goal of this interventional study is to see if the daily use of red light therapy called photobiomodulation can help sore skin and sore mouths in children having radiotherapy.

All children aged 0-16 years old who are receiving either proton or photon radiotherapy treatment, except to the brain only, will be asked if they would like to join the study.

The main questions it aims to answer are:

1. Does the use of red light therapy help the skin side effects in children and young people undergoing proton or photon therapy?
2. Does the use of red light therapy help the mouth side effects in children and young people undergoing proton or photon therapy in the head and neck area?

Researchers will compare the patients enrolled on to the study with a like for like historic patient to see if red light therapy improves the sore skin and sore mouths caused by proton or photon therapy.

Participants will have a daily treatment with red light therapy alongside their daily proton or photon treatment fraction.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patient receiving a treatment course of either proton or photon therapy - Craniospinal treatment field, Head and Neck treatment fields and body treatment fields.

Exclusion Criteria:

* Paediatric patients receiving focal brain only proton or photon radiotherapy.
* Paediatric patients receiving a single fraction of proton or photon therapy.
* Total Body Irradiation patients.

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 248 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Paediatric Participants with Treatment-Related Skin Toxicity as Assessed by RTOG | The participant will be assessed from day one until the end of their proton or photon radiotherapy treatment course, up to 8 weeks.
  RTOG Skin Toxicity score range:
  Grade 0: no change Grade 1: dull erythema, decreased sweating Grade 2: moderate oedema, bright erythema, pitting oedema Grade 3: confluent moist desquamation, pitting oedema Grade 4: Ulceration, haemorrhage and necrosis.

SECONDARY OUTCOMES:
Number of Head and Neck Participants with Treatment-Related Mucositis as Assessed by CTCAE v4.0 | The participant will be assessed from day one until the end of their proton or photon radiotherapy treatment course, up to 8 weeks.
  CTCAE mucositis scoring scale:
  Grade 0: No mucositis. Grade 1: Asymptomatic or mild symptoms; intervention not indicated. Grade 2: Moderate pain or ulcer that does not interfere with oral intake; modified diet indicated.
  Grade 3: Severe pain; interfering with oral intake. Grade 4: Life-threatening consequences; urgent intervention indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Ed Smith, Study Director — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robijns J, Lodewijckx J, Claes S, Van Bever L, Pannekoeke L, Censabella S, Busse L, Colson D, Kaminski I, Broux V, Puts S, Vanmechelen S, Timmermans A, Noe L, Bulens P, Govers M, Maes A, Mebis J. Photobiomodulation therapy for the prevention of acute radiation dermatitis in head and neck cancer patients (DERMISHEAD trial). Radiother Oncol. 2021 May;158:268-275. doi: 10.1016/j.radonc.2021.03.002. Epub 2021 Mar 10. PMID 33711412
- [Background] Heggie C, Gray-Burrows KA, Day PF, Phillips B. An exploration of the use of photobiomodulation for management of oral mucositis in children and young people undergoing cancer treatment in the UK. Support Care Cancer. 2022 Dec;30(12):10179-10190. doi: 10.1007/s00520-022-07450-3. Epub 2022 Nov 9. PMID 36350380
- [Background] Gobbo M, Rico V, Marta GN, Caini S, Ryan Wolf J, van den Hurk C, Beveridge M, Lam H, Bonomo P, Chow E, Behroozian T. Photobiomodulation therapy for the prevention of acute radiation dermatitis: a systematic review and meta-analysis. Support Care Cancer. 2023 Mar 23;31(4):227. doi: 10.1007/s00520-023-07673-y. PMID 36952036
- [Background] Bensadoun RJ, Epstein JB, Nair RG, Barasch A, Raber-Durlacher JE, Migliorati C, Genot-Klastersky MT, Treister N, Arany P, Lodewijckx J, Robijns J; World Association for Laser Therapy (WALT). Safety and efficacy of photobiomodulation therapy in oncology: A systematic review. Cancer Med. 2020 Nov;9(22):8279-8300. doi: 10.1002/cam4.3582. Epub 2020 Oct 26. PMID 33107198